CLINICAL TRIAL: NCT02433418
Title: Tubal Flushing Using Water Soluble Media for Unexplained Infertility: A Randomized Controlled Trial
Brief Title: Tubal Flushing Using Water Soluble Media for Unexplained Infertility
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sub 9
Record Dates: First submitted 2015-04-24; First posted 2015-05-05 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tubal flushing with Urografin® (Active Comparator): Women will have HSG using water soluble media
  Interventions: Procedure: Tubal flushing by Urografin®; Drug: Diclofenac
- Control group (No Intervention): Women will not receive any intervention

INTERVENTIONS:
Procedure: Tubal flushing by Urografin® — Women will have tubal flushing through HSG using water soluble media (Urographin ®)
  Arms: Tubal flushing with Urografin®
Drug: Diclofenac — Women will receive oral diclofenac 50 mg (voltaren ®) 1 hour before hysterosalpingography
  Arms: Tubal flushing with Urografin®

SUMMARY:
300 women with unexplained infertility will be randomly divided into 2 equal groups: Group 1 will be offered tubal flushing with water soluble media through hysterosalpingography (HSG) and group 2 will receive no intervention

DETAILED DESCRIPTION:
The potential therapeutic effect of diagnostic tubal patency testing has been debated for over 40 years. Tubal flushing might involve water- or oil-soluble media. Current practice usually involves water-soluble media when tubal flushing is performed at laparoscopy. A systematic review showed a significant increase in pregnancy rates with tubal flushing using oil-soluble contrast media when compared with no treatment. Tubal flushing with oil soluble contrast media was associated with an increase in the odds of live birth when compared with tubal flushing with water-soluble media. There were no trials assessing tubal flushing with water-soluble media versus no treatment. The potential consequences of extravasations of oil-soluble contrast media into the pelvic cavity and fallopian tubes may be associated with anaphylaxis and lipogranuloma. It has been reported that Further randomised controlled trials are needed to evaluate the potentially therapeutic effects of tubal flushing with water-soluble media.

All patients attending the subfertility clinic with infertility, normal semen analysis and evidence of ovulation will be invited to participate in the study. The nature of the study and its expected values will be explained and only women who provide written consents will be included in the study.

Three hundred women will be divided into 2 equal groups using computer generated random numbers: Group 1 will have tubal flushing with HSG using water soluble media and group 2 will be the control group receiving no intervention.

Women undergoing HSG will be given 50 mg of diclofenac (Voltaren® Novartis) 1 hour before the procedure. The HSG will be performed in the same room, on the same table and with the same technique to maintain consistency and limit confounding variables.

The HSG procedure will performed in a lithotomy position. A sterile metal speculum was used to visualize the uterine cervix. Antiseptic solution will be used to wash the vagina and cervix. A single-toothed tenaculum will be placed on the anterior lip of the cervix. A metal cannula will be gently inserted into the external cervical os, the cannula and tenaculum will be secured together, and the speculum will be removed. Gentle traction will be placed on the tenaculum, and 15 mL to 20 mL of water-soluble media (Sodium Amidotrizoate; urografin®, Bayer, Germany) will be instilled slowly via the cannula to prevent pain while the necessary images were obtained. After the procedure, the instruments will be removed and the patient will be observed for 30 minutes.

Women will be followed up monthly for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* infertility for one year
* Normal semen analysis
* Normal ovulation

Exclusion Criteria:

* Allergy to Iodine
* Metformin therapy
* Tubal block

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy | Monthly, up to 12 months
  Pregnancy will be defined as the presence of an intrauterine sac by vaginal ultrasound

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - BeniSuef University hospitals, BeniSuef
  - Cairo University Hospitals, Cairo

REFERENCES:
- [Background] Steiner AZ, Meyer WR, Clark RL, Hartmann KE. Oil-soluble contrast during hysterosalpingography in women with proven tubal patency. Obstet Gynecol. 2003 Jan;101(1):109-13. doi: 10.1016/s0029-7844(02)02390-6. PMID 12517654
- [Background] Spring DB, Barkan HE, Pruyn SC. Potential therapeutic effects of contrast materials in hysterosalpingography: a prospective randomized clinical trial. Kaiser Permanente Infertility Work Group. Radiology. 2000 Jan;214(1):53-7. doi: 10.1148/radiology.214.1.r00ja2353. PMID 10644101
- [Background] Luttjeboer F, Harada T, Hughes E, Johnson N, Lilford R, Mol BW. Tubal flushing for subfertility. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD003718. doi: 10.1002/14651858.CD003718.pub3. PMID 17636730
- [Derived] Wang R, Watson A, Johnson N, Cheung K, Fitzgerald C, Mol BWJ, Mohiyiddeen L. Tubal flushing for subfertility. Cochrane Database Syst Rev. 2020 Oct 15;10(10):CD003718. doi: 10.1002/14651858.CD003718.pub5. PMID 33053612